CLINICAL TRIAL: NCT06293118
Title: The Chronic Effect of Ischemic Conditioning on Motor Function, Cognitive Performance, and Immune System in Individuals with Parkinson's Disease
Brief Title: The Effects of Ischemic Conditioning in Individuals with Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Unifesp Escola Paulista de Medicina (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 71055423.3.0000.0071
Record Dates: First submitted 2024-02-19; First posted 2024-03-05 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease
Keywords: ischemic conditioning; immune system; motor function; cognitive performance; Parkinson disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: 1. Ischemic conditioning group
  2. control group (Sham)
Who Masked: Participant
Masking Description: Patients were unaware of the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Ischemic conditioning group (Experimental): Therapy will be performed bilaterally on the upper limbs. The ischemic conditioning group will perform 4 times, 8 cycles with 30 seconds of ischemia (80 - 200 mmHg) with 5 seconds of reperfusion in each cycle. Ischemia cycles are controlled by a device (KAATSU C3 - KAATSU GLOBAL / USA) In the first cycle, participants will be subjected to pressures of 80 to 150 mmHg. In the 3 subsequent cycles, pressures from 130 to 200 mmHg will be applied.
  Interventions: Device: Ischemic conditioning group
- Sham group (Sham Comparator): Participants in the control group (Sham) will perform 4 cycles of 5 minutes of ischemia (30 mmHg) with 4 subsequent cycles of reperfusion (rest) bilaterally in the arms with a sphygmomanometer (Welch Allyn DS44-11BR Durashock).
  Interventions: Device: Sham group

INTERVENTIONS:
Device: Ischemic conditioning group — The ischemic conditioning protocol will consist of a period of 12 weeks (24 sessions) with a frequency of 2 weekly sessions lasting between 15 and 20 minutes each. Therapy will be performed bilaterally on the upper limbs. The ischemic conditioning group will perform 4 times, 8 cycles with 30 seconds of ischemia (80 - 200 mmHg) with 5 seconds of reperfusion in each cycle. Ischemia cycles are controlled by a device (KAATSU C3 - KAATSU GLOBAL / USA) with customized ischemia programs, partially restricting blood flow through special pressure cuffs that are internally valved, providing greater comfort and safety for these patients who typically have stiffness in the affected limb and localized muscle pain. In the first cycle, participants will be subjected to pressures of 80 to 150 mmHg. In the 3 subsequent cycles, pressures from 130 to 200 mmHg will be applied.
  Arms: Ischemic conditioning group
Device: Sham group — Participants in the control group (Sham) will perform 4 cycles of 5 minutes of ischemia (30 mmHg) with 4 subsequent cycles of reperfusion (rest) bilaterally in the arms with a sphygmomanometer
  Arms: Sham group

SUMMARY:
Ischemic conditioning (IC) is a promising therapy that can mimic the physiological effects of physical exercise. IC consists of using a cuff to measure blood pressure and calibrate 200 mmHg on the upper or lower limb. Thus, at alternating intervals of 5 minutes, ischemia or reperfusion occurs, depending on whether the cuff is inflated or deflated. IC induces changes in spinal cord excitability for the last reflex reactions of recruited motoneurons with improved balance control in healthy young people and improved learning in the elderly. The objective of the present study is to evaluate the chronic effect of IC on the motor function and cognitive performance of patients with Parkinson's disease. Furthermore, the investigators will evaluate secondary outcomes such as mobility, quality of life, and immunological responses.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disorder that causes a variety of motor and non-motor symptoms. Typically, patients with PD suffer from disabilities and secondary complications even when the disease is optimally treated, and many patients still have sedentary lifestyles, which in turn result in higher rates of mortality and comorbidity. Physical activity is an essential element in maintaining daily functional capabilities and quality of life. However, patients with PD have motor and non-motor deficits that can prevent or limit physical exercise, such as running or resistance exercise. Ischemic conditioning (IC) is a promising therapy that can mimic the physiological effects of physical exercise. IC consists of using a cuff to measure blood pressure, calibrated between 180 and 200 mmHg on the upper or lower limb. Thus, at alternating intervals of 5 minutes, ischemia or reperfusion occurs, depending on whether the cuff is inflated or deflated. IC induces changes in spinal cord excitability for the last reflex reactions of recruited motoneurons with improved balance control in healthy young people and improved learning in the elderly. Recently, IC has been shown to improve cognitive performance in neurological patients with stroke, subcortical ischemia, and vascular dementia. However, there are no studies that have evaluated the effect of IC on motor and cognitive performance in patients with PD. The objective of the present study is to evaluate the chronic effect of IC on the motor and cognitive performance of patients with PD. Furthermore, the investigators intend to evaluate other secondary outcomes such as mobility, quality of life, and immunological responses.

ELIGIBILITY:
Inclusion Criteria:

* PD patients aged 40 years or older;
* Diagnosis of PD without cognitive complaints or with complaints, but without impact on daily activities;

Exclusion Criteria:

* Patients with uncontrolled diabetes mellitus or peripheral neuropathy;
* Uncontrolled arterial hypertension (BP>160/100mmHg);
* Uncontrolled diabetes (Fasting glucose > 250mg/dl, peripheral retinopathy or diabetic ketoacidosis);
* Uncontrolled dyslipidemia (total chol > 220mg/dL);
* Pre-existing autoimmune diseases;
* Infectious conditions for less than 1 month;
* Neurological problems that prevent training from being carried out;
* History of anemia, cerebral vascular disease, myocardial infarction in the last 6 months;
* Previous deep vein thrombosis;
* Smoking < 6 months;
* Symptomatic peripheral arterial obstructive disease;
* Cognitive dysfunction: Moca < 24.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale | Before intervention and at week 12
  0-260 points: A higher score indicates greater impairment
Montreal cognitive assesment | Before intervention and at week 12
  Maximum score: 30 points; Normal cognition: 26-30 points; Mild cognitive impairment (MCI): Below 26 points

SECONDARY OUTCOMES:
The Parkinson's Disease Questionnaire-39 | Before intervention and at week 12
  The overall score ranges from 0 to 100%, with higher scores indicating a greater negative impact of Parkinson's Disease on the patient's quality of life.
Timed up and go | Before intervention and at week 12
  <10 seconds: Individuals are generally able to perform most daily activities independently without assistance; 10-19 seconds: Indicates independence in most daily activities but may suggest slight mobility limitations; 20-29 seconds: Suggests the need for assistance with mobility, especially for more challenging tasks;
  ≥30 seconds: Indicates a high fall risk, and the individual likely needs assistance with many daily tasks and may require mobility aids.
Assessment of cellular and soluble immune response | Before intervention and at week 12
  The patient's peripheral blood will be collected in three EDTA tubes of 5 mL each before and after 12 weeks of application of the ischemic conditioning protocol. From the blood samples, plasma will be obtained for quantification of soluble mediators, followed by the isolation/storage of peripheral blood mononuclear cells (PBMC or Peripheral Blood Mononuclear Cell) for phenotypic characterization of subpopulations of T and B lymphocytes, NK cells, myeloids and monocytes
Quantifications of systemic soluble mediators | Before intervention and at week 12
  Initially, the EDTA tubes containing the blood will be centrifuged for 5 minutes at 400 x g and 20 ºC to separate the plasma. The collected plasma will be aliquoted into cryotubes and stored at -80ºC until the tests are carried out. Quantification of systemic soluble mediators will be performed using the MILLIPLEX® Human Cytokine/Chemokine/Growth Factor Panel A Kit H - Immunology Multiplex Assay (Merck Millipore, Massachusetts, USA). The panel of analytes included chemokines, growth factors, pro-inflammatory cytokines and regulatory cytokines: FGF-2/FGF-basic, G-CSF, GM-CSF, IFNa2,IFNy, IL-1a, IL-1b, IL-1RA , IL-2, IL-4, IL-6, IL-7, IL-8/CXCL8, IL-10, IL-12 (p40), IL-12 (p70), IL-13, IL-15, IL -17A/CTLA8, IL-18, IP-10/CXCL10, MCP-1/CCL2, MCP-3/CCL7, M-CSF, MIG/CXCL9, MIP-1a/CCL3, MIP-1b/CCL4, PDGF-AB /BB, RANTES/CCL5, TNFa, TNFb/Lymphotoxin-a, VEGF-A, HIF-1ą. The PCR, BNDF, and Irisin proteins will be measured using single-plex assays.
PBMC acquisition and flow cytometry | Before intervention and at week 12
  Finally, a minimum of 100,000 events will be acquired on the BD LSRFortessa™ flow cytometer (BD Biosciences).

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Gollob, PhD, Principal Investigator — Hospital Israelita Albert Einstein

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poewe et al. Parkinson disease. Nat Rev 2017;3:1-21. doi:10.1038/nrdp.2017.13
- [Background] Dickson DW, Braak H, Duda JE, Duyckaerts C, Gasser T, Halliday GM, Hardy J, Leverenz JB, Del Tredici K, Wszolek ZK, Litvan I. Neuropathological assessment of Parkinson's disease: refining the diagnostic criteria. Lancet Neurol. 2009 Dec;8(12):1150-7. doi: 10.1016/S1474-4422(09)70238-8. PMID 19909913
- [Background] Kaushik S, Cuervo AM. Proteostasis and aging. Nat Med. 2015 Dec;21(12):1406-15. doi: 10.1038/nm.4001. PMID 26646497
- [Background] Bose A, Beal MF. Mitochondrial dysfunction in Parkinson's disease. J Neurochem. 2016 Oct;139 Suppl 1:216-231. doi: 10.1111/jnc.13731. Epub 2016 Aug 21. PMID 27546335
- [Background] Poewe W. Clinical measures of progression in Parkinson's disease. Mov Disord. 2009;24 Suppl 2:S671-6. doi: 10.1002/mds.22600. PMID 19877235
- [Background] Post B, Merkus MP, de Bie RM, de Haan RJ, Speelman JD. Unified Parkinson's disease rating scale motor examination: are ratings of nurses, residents in neurology, and movement disorders specialists interchangeable? Mov Disord. 2005 Dec;20(12):1577-84. doi: 10.1002/mds.20640. PMID 16116612
- [Background] Schapira AHV, Chaudhuri KR, Jenner P. Non-motor features of Parkinson disease. Nat Rev Neurosci. 2017 Jul;18(7):435-450. doi: 10.1038/nrn.2017.62. Epub 2017 Jun 8. PMID 28592904
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Xu R, He Q, Wang Y, Yang Y, Guo ZN. Therapeutic Potential of Remote Ischemic Conditioning in Vascular Cognitive Impairment. Front Cell Neurosci. 2021 Aug 3;15:706759. doi: 10.3389/fncel.2021.706759. eCollection 2021. PMID 34413726
- [Background] Loukogeorgakis SP, Williams R, Panagiotidou AT, Kolvekar SK, Donald A, Cole TJ, Yellon DM, Deanfield JE, MacAllister RJ. Transient limb ischemia induces remote preconditioning and remote postconditioning in humans by a K(ATP)-channel dependent mechanism. Circulation. 2007 Sep 18;116(12):1386-95. doi: 10.1161/CIRCULATIONAHA.106.653782. Epub 2007 Aug 27. PMID 17724264
- [Background] Strijdom H, Friedrich SO, Hattingh S, Chamane N, Lochner A. Hypoxia-induced regulation of nitric oxide synthase in cardiac endothelial cells and myocytes and the role of the PI3-K/PKB pathway. Mol Cell Biochem. 2009 Jan;321(1-2):23-35. doi: 10.1007/s11010-008-9906-2. Epub 2008 Sep 14. PMID 18791856
- [Background] Sutter EN, Mattlage AE, Bland MD, Cherry-Allen KM, Harrison E, Surkar SM, Gidday JM, Chen L, Hershey T, Lee JM, Lang CE. Remote Limb Ischemic Conditioning and Motor Learning: Evaluation of Factors Influencing Response in Older Adults. Transl Stroke Res. 2019 Aug;10(4):362-371. doi: 10.1007/s12975-018-0653-8. Epub 2018 Aug 7. PMID 30088217
- [Background] Guo ZN, Guo WT, Liu J, Chang J, Ma H, Zhang P, Zhang FL, Han K, Hu HH, Jin H, Sun X, Simpson DM, Yang Y. Changes in cerebral autoregulation and blood biomarkers after remote ischemic preconditioning. Neurology. 2019 Jul 2;93(1):e8-e19. doi: 10.1212/WNL.0000000000007732. Epub 2019 May 29. PMID 31142636
- [Background] He Z, Xu N, Qi S. Remote ischemic preconditioning improves the cognitive function of elderly patients following colon surgery: A randomized clinical trial. Medicine (Baltimore). 2017 Apr;96(17):e6719. doi: 10.1097/MD.0000000000006719. PMID 28445286
- [Background] Zhou D, Ding J, Ya J, Pan L, Bai C, Guan J, Wang Z, Jin K, Yang Q, Ji X, Meng R. Efficacy of remote ischemic conditioning on improving WMHs and cognition in very elderly patients with intracranial atherosclerotic stenosis. Aging (Albany NY). 2019 Jan 28;11(2):634-648. doi: 10.18632/aging.101764. PMID 30689549
- [Background] Liao Z, Bu Y, Li M, Han R, Zhang N, Hao J, Jiang W. Remote ischemic conditioning improves cognition in patients with subcortical ischemic vascular dementia. BMC Neurol. 2019 Aug 23;19(1):206. doi: 10.1186/s12883-019-1435-y. PMID 31443692
- [Background] Movement Disorder Society Task Force on Rating Scales for Parkinson's Disease. The Unified Parkinson's Disease Rating Scale (UPDRS): status and recommendations. Mov Disord. 2003 Jul;18(7):738-50. doi: 10.1002/mds.10473. PMID 12815652